CLINICAL TRIAL: NCT03024879
Title: Influence of Erythromycin on ad Libitum Food Intake and the Evaluation of Motilin in Food Timing in Healthy Volunteers and Patients
Brief Title: The Effect of Motilin on the Frequency and Amount of Food Intake
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MotilinAndFoodIntake
Record Dates: First submitted 2016-05-23; First posted 2017-01-19 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Obesity
Keywords: Motilin; Erythromycin; Food intake
MeSH Terms: conditions — Obesity | interventions — Erythromycin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythromycin (Active Comparator): 40 mg of erythromycin will be administered intravenously over a period of 20 min in a saline solution of 100 ml
  Interventions: Drug: Erythromycin
- Placebo (Placebo Comparator): a saline solution of 100 ml will be administered intravenously over a period of 20 min
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Erythromycin
  Arms: Erythromycin
Drug: Saline
  Arms: Placebo

SUMMARY:
In this study, the investigators aimed at evaluating the role of motilin in the regulation of food intake. Motilin, a gastrointestinal hormone, is a hunger signal in healthy volunteers and is significantly increased in obese patients. Its role in food intake regulation might contribute to the pathogenesis of obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m² for lean volunteers
* BMI > 30 kg/m² for obese volunteers
* Subject is capable and willing to give informed consent
* Female volunteers of child bearing potential must use oral, injected or implanted hormonal methods of contraception

Exclusion Criteria:

* Female volunteer is pregnant or breastfeeding
* GI diseases, major abdominal surgery
* Major psychiatric illnesses
* Volunteers that use drugs affecting the GI tract or the central nervous system
* Volunteers suffering from endocrine diseases such as diabetes, Cushing's disease, Addison's disease, hypothalamic tumor
* Volunteers that have undergone surgical procedure for weight loss

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in food intake, assessed by caloric intake, after intravenous administration of erythromycin compared to placebo | Caloric intake will be assessed 1 hour after the start of infusion and the start of ad libitum food intake

SECONDARY OUTCOMES:
Frequency of food intake correlated with motilin plasma levels | Assessment will be done over a period of 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deloose E, Biesiekierski JR, Vanheel H, Depoortere I, Tack J. Effect of motilin receptor activation on food intake and food timing. Am J Clin Nutr. 2018 Apr 1;107(4):537-543. doi: 10.1093/ajcn/nqx044. PMID 29635488